CLINICAL TRIAL: NCT00513981
Title: Study to Determine the Maximum Tolerated Time of Infusion for High-Dose Methotrexate, Administered as a Continuous Intravenous Infusion at a Dose of 6g/m² Per 24 Hours of Infusion Time
Brief Title: High-Dose Methotrexate in Treating Young Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-NAG-2005-13; CDR0000560133 (Registry Identifier: PDQ (Physician Data Query)); EU-20744; EUDRACT-2005-001757-13
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; recurrent osteosarcoma; recurrent childhood soft tissue sarcoma; recurrent childhood ependymoma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Sarcoma; Osteosarcoma; Familial ependymoma | interventions — Leucovorin; Methotrexate; Mass Spectrometry

INTERVENTIONS:
Drug: leucovorin calcium
Drug: methotrexate
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as high-dose methotrexate work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoprotective drugs, such as leucovorin calcium, may protect normal cells from the side effects of chemotherapy.

PURPOSE: This phase I trial is studying the side effects, best way to give, and best dose of high-dose methotrexate in treating patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated time to exposure to high-dose methotrexate when administered as a continuous infusion at a dose of 6 g/m² per 24 hours.
* To relate the methotrexate schedules investigated to the magnitude and duration of changes in plasma homocysteine and methionine.
* To relate evidence of the systemic effect of methotrexate through changes in plasma homocysteine and methionine to any hepatic, neurological, or antiproliferative toxicity observed in the study group.

OUTLINE: Patients receive a continuous infusion of high-dose methotrexate IV over 24, 30, 36, or 42 hours depending on time of study entry. Beginning at hour 42 or 48, patients receive leucovorin calcium IV every 6 hours for 3 days or until plasma methotrexate concentration is < 0.2 µM. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study and analyzed for pharmacodynamic effects on plasma homocysteine and methionine by gas chromatography/mass spectrometry techniques.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignancy, including but not limited to, any of the following:

  * Patients with MRI findings in keeping with a diffuse intrinsic pontine glioma will be eligible without histological confirmation of tumor type

    * Patients with a diagnosis of diffuse intrinsic pontine glioma who are not eligible for the erlotinib hydrochloride phase I study (CCLG-NAG-2005-09)
  * Patients with relapsed ependymoma following the CCLG phase II study of intravenous etoposide (CCLG-CNS-2001-4) or prior to this are eligible at the discretion of the physician
  * Patients with relapsed osteogenic sarcoma, other soft tissue sarcomas, or other solid tumors may be suitable for this study at the discretion of the physician
* Radiologically evaluable disease without bone marrow involvement

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Lansky performance status (PS) 30-100% (for patients ≤ 12 years of age)
* ECOG PS ≤ 2 (for patients ≥ 13 years of age)
* Life expectancy ≥ 9 weeks
* ANC > 1,000/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 9 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN) for age
* Serum total bilirubin normal
* AST or ALT ≤ 2 times ULN
* Glomerular filtration rate ≥ 60 mL/min
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Poor medical risk because of nonmalignant systemic disease or uncontrolled infection
* Concurrent malignancies at other sites

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Prophylactic trimethoprim-sulfamethoxazole must be stopped 1 week prior to methotrexate administration

Exclusion criteria:

* Received chemotherapy or biologic therapy within the past 4 weeks
* Received radiotherapy within the past 6 weeks

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated infusion time for high-dose methotrexate

SECONDARY OUTCOMES:
Plasma biochemical evidence of the systemic effect of methotrexate in terms of changes in plasma homocysteine and methionine

CONTACTS AND LOCATIONS:
Overall Officials: Eddy J. Estlin, Principal Investigator — Royal Manchester Children's Hospital
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - University College Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales